CLINICAL TRIAL: NCT01001689
Title: Fit For Delivery: A Study of the Effect of Exercise Intervention and Nutritional Counselling on Pregnancy Outcome.
Brief Title: Fit For Delivery: A Study of the Effect of Exercise Sessions and Nutritional Counselling on Pregnancy Outcome
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 811363
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy; Obesity; Diabetes
Keywords: Pregnancy; Preventive health care; Fitness; Nutrition; Obesity; Diabetes; Weight gain
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Gain | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional counseling + exercise groups (Experimental): Women in this arm will receive 2 telephone consultations on nutritional health during pregnancy, be invited to 2 evening meetings with nutritional topics and have access to a password protected internet site with topics related to nutrition and fitness in pregnancy. They will also be enrolled in an exercise group which will meet twice weekly, and be encouraged to exercise on their own 1-2 times each week.
  Interventions: Behavioral: Nutritional counseling + exercise groups
- control (No Intervention): Women in this arm of the study will receive routine pregnancy care.

INTERVENTIONS:
Behavioral: Nutritional counseling + exercise groups — Two telephone consultations on nutritional topics and twice weekly exercise groups. Access to a password-protected internet site with information on healthy lifestyle during pregnancy. Two evening meetings with information on healthy pregnancy lifestyle.
  Arms: Nutritional counseling + exercise groups

SUMMARY:
"Fit for Delivery" is a randomized, controlled study to examine the effects of an intervention during pregnancy which consists of exercise groups and nutritional counselling. The investigators will assess the outcomes of gestational weight gain, postpartum weight retention, large newborns, glucose regulation, and the incidence of complications of pregnancy and delivery such as gestational diabetes and Cesarean section.

DETAILED DESCRIPTION:
"Fit for Delivery" is a randomized, controlled study to examine the effects of an intervention during pregnancy which consists of exercise groups and nutritional counselling. The investigators intend to study 600 women who are expecting their first child, and include them in the study at the time of their first appointment at their local healthcare clinic, when they are between 12 and 20 weeks of pregnancy. All women who wish to participate will sign an informed consent.

Women who are randomly assigned to the intervention group will receive two telephone consultations with nutritional advice on healthy eating during pregnancy. They will also be counselled about appropriate weight gain during pregnancy given their pre-pregnancy body mass index. They will be assigned to an exercise group which will meet twice a week for a specially designed workout, and will be encouraged to exercise once or twice weekly on their own. Women in the intervention group will also have access to a password-protected internet site with information on healthy living during pregnancy, and be invited to 2 or 3 evening classes with nutritional information. Women who are randomly assigned to the control group will receive routine pregnancy care.

All women in the study will be studied using:

* questionaires
* two ultrasound examinations (at 30 and 36 weeks of pregnancy),
* blood tests, including a 2 hour glucose challenge test, and measurement of hormones which regulate blood glucose levels
* weighing of the participant, including use of a bioimpedance scale
* weighing and measuring of her newborn baby,
* blood tests from the umbilical cord, measuring hormones which regulate blood glucose levels
* review of hospital records regarding mode of delivery, delivery complications and possible neonatal admissions for the newborn child.

The investigators' hypothesis is that an intervention in the form of nutritional information and exercise groups will:

1. Affect the amount of weight women gain in pregnancy, and the amount of weight they retain 12 month after delivery
2. Affect the percentage of newborns who have a birthweight over 4 kilo, or who have a birthweight at or above the 90th percentile for Norwegian newborns.
3. Affect the blood sugar level and the incidence of gestational diabetes.
4. Affect the incidence of operative deliveries and the delivery by Cesarean section.
5. Affect the serum concentrations of hormones regulating blood sugar levels, measured in both participants and their newborns.

ELIGIBILITY:
Inclusion Criteria:

* Expecting first child
* Gestational weeks 12-20
* Residence in one of the following towns: Kristiansand, Søgne, Sogndalen, Vennesla, Lillesand, Mandal

Exclusion Criteria:

* Twin or other multiple pregnancy
* Preexisting diabetes
* Physical handicap which precludes participation in exercise groups
* Ongoing drug addiction
* Serious mental disorder
* BMI at or below 19 before pregnancy
* Inability to read/write Norwegian or English

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain in pregnancy | Measured at the time of delivery
  weight gain in kg
Weight of the newborn | Measured at the time of delivery
  weight in grams at delivery
Maternal fasting serum glucose level | Measured at gestational week 30
  serum glucose
Incidence of operative delivery, both cesarean section and operative vaginal delivery | Assessed following delivery
  number of participants delivered by operative vaginal or cesarean section
Maternal body composition | Measured at 36 weeks of gestation
  Measured using bioimpedance scale

SECONDARY OUTCOMES:
Maternal weight retention | 12 months after delivery
  weight change in kg from pre-pregnancy weight
Measurement of serum levels of hormones which regulate serum glucose levels, in both the pregnant woman and her newborn baby. | Mother measured at gestational week 30, baby measured at delivery
  insulin, leptin
Incidence of women with serum glucose levels >7.8 mmol/l after 2 hour glucose challenge test | Assessed at gestational week 30
  results of glucose challege test
Incidence of delivery complications | Assessed following delivery
  incidence of third and fourth degree tearing, hemmorhage
Proportion of newborns with birth weight over the 90th percentile for gestational age | Assessed following delivery
  weight at gestation, adjusted for population characteristics stratified by sex and gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Vistad, MD, PhD, Principal Investigator — Sorland Hospital HF; Tore Henriksen, MD, PhD, Study Chair — University Hospital of Oslo, Rikshospital
Locations (1):
- Sorlandet Hospital, Kristiansand, Vest Agder, Norway

REFERENCES:
- [Background] Sagedal LR, Overby NC, Bere E, Torstveit MK, Lohne-Seiler H, Smastuen M, Hillesund ER, Henriksen T, Vistad I. Lifestyle intervention to limit gestational weight gain: the Norwegian Fit for Delivery randomised controlled trial. BJOG. 2017 Jan;124(1):97-109. doi: 10.1111/1471-0528.13862. Epub 2016 Jan 14. PMID 26768233
- [Background] Sagedal LR, Sanda B, Overby NC, Bere E, Torstveit MK, Lohne-Seiler H, Hillesund ER, Pripp AH, Henriksen T, Vistad I. The effect of prenatal lifestyle intervention on weight retention 12 months postpartum: results of the Norwegian Fit for Delivery randomised controlled trial. BJOG. 2017 Jan;124(1):111-121. doi: 10.1111/1471-0528.13863. Epub 2016 Jan 20. PMID 26786294
- [Derived] Hillesund ER, Seland S, Bere E, Sagedal LR, Torstveit MK, Lohne-Seiler H, Vistad I, Overby NC. Preeclampsia and gestational weight gain in the Norwegian Fit for Delivery trial. BMC Res Notes. 2018 May 8;11(1):282. doi: 10.1186/s13104-018-3396-4. PMID 29739447
- [Derived] Haakstad LAH, Vistad I, Sagedal LR, Lohne-Seiler H, Torstveit MK. How does a lifestyle intervention during pregnancy influence perceived barriers to leisure-time physical activity? The Norwegian fit for delivery study, a randomized controlled trial. BMC Pregnancy Childbirth. 2018 May 3;18(1):127. doi: 10.1186/s12884-018-1771-8. PMID 29724165
- [Derived] Sagedal LR, Vistad I, Overby NC, Bere E, Torstveit MK, Lohne-Seiler H, Hillesund ER, Pripp A, Henriksen T. The effect of a prenatal lifestyle intervention on glucose metabolism: results of the Norwegian Fit for Delivery randomized controlled trial. BMC Pregnancy Childbirth. 2017 Jun 2;17(1):167. doi: 10.1186/s12884-017-1340-6. PMID 28577545
- [Derived] Skreden M, Bere E, Sagedal LR, Vistad I, Overby NC. Changes in fruit and vegetable consumption habits from pre-pregnancy to early pregnancy among Norwegian women. BMC Pregnancy Childbirth. 2017 Apr 4;17(1):107. doi: 10.1186/s12884-017-1291-y. PMID 28376732
- [Derived] Sagedal LR, Overby NC, Lohne-Seiler H, Bere E, Torstveit MK, Henriksen T, Vistad I. Study protocol: fit for delivery - can a lifestyle intervention in pregnancy result in measurable health benefits for mothers and newborns? A randomized controlled trial. BMC Public Health. 2013 Feb 13;13:132. doi: 10.1186/1471-2458-13-132. PMID 23406306